CLINICAL TRIAL: NCT05521425
Title: Efficacy and Safety of "Helping Hands": A 3D Printed Device of Peritoneal Dialysis Adopted in Continuous Ambulatory Peritoneal Dialysis: A Randomized Controlled Trial
Brief Title: Randomized Controlled Trial on 3D Printed Assistive Device for Continuous Ambulatory Peritoneal Dialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Elizabeth Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Carina Ho, Principal Investigator, Queen Elizabeth Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-0266-FR-1
Record Dates: First submitted 2022-08-22; First posted 2022-08-30 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Renal Failure Chronic
Keywords: Continuous Ambulatory Peritoneal Dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Non-inferiority, Paralleled, Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: After completion of written consent, participants were randomly assigned to either intervention or control group. Outcomes assessors (and facilitators for phone interview for follow-up action) were independent, not knowing the condition of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Training + "Helping Hands" provided for CAPD bag exchange procedures at home
  Interventions: Device: "Helping Hands" for CAPD bag exchange procedures
- Control Group (No Intervention): Training alone (without "Helping Hands" provided to assist in bag exchange procedures)

INTERVENTIONS:
Device: "Helping Hands" for CAPD bag exchange procedures — Training served as "Treatment As Usual" (TAU) for all participants; The difference between two groups was whether "Helping hands" were provided to participants for CAPD bag exchange procedures at home.
  Arms: Intervention Group

SUMMARY:
Touch contamination during bag exchange in Continuous Ambulatory Peritoneal Dialysis (CAPD) is a common cause of CAPD-related peritonitis. An innovative 3D-printed assistive device "Helping Hands" was designed to minimize direct touch of tubing during CAPD bag exchange to allow a safer connection process for patients with Chronic Kidney Disease (CKD) to reduce the risk of CAPD-related peritonitis. Through this randomized control, the investigators aimed to evaluate the safety and efficacy of "Helping Hands" in CAPD bag exchange procedure for patients on CAPD therapy.

DETAILED DESCRIPTION:
The study will be conducted in the Renal Unit, Queen Elizabeth Hospital (QEH). All new CAPD patients using Ultrabag Peritoneal Dialysis (PD) system will be screened and invited to participate in this study by occupational therapist or nurse. Patients with cognitive impairment, psychiatric illness, acute illness that requires frequent hospital admissions (>3 episodes with hospital stay over 1 week), or current adoption of other type of assistive device in CAPD bag exchange will be excluded. Eligible patients will be randomly allocated to either intervention group (using "Helping Hands") or control group. Participants in both arms will receive a standard 5-day CAPD training program and then perform a competency test for bag exchange conducted by an independent Advanced Practice Nurses. Irrespective of grouping, participants will receive brief phone interviews by clerks (who did not take the role as investigators) from the QEH Renal Unit with two sets of questionnaire measuring their health related conditions at 4 time points i) A0 (baseline); ii) A1 (last day of CAPD training); iii) A2 (4-month post-training follow-up); and iv) A3 (8-month post-training follow-up). Intervention group will receive additional training on using "Helping Hands" as assistive device in performing bag exchange and will have extra follow-up assessment at the 4th and 8th month post-training to ensure their competence in using "Helping Hands" device to perform CAPD exchanges. Relevant clinical data, such as peritonitis record, will be collected during their routine follow-up in the dialysis center or by clinical medical system.

This is a non-inferiority study with the objective of establishing the safety and efficacy of "Helping hands" device for patients doing CAPD bag exchanges using UltraBag PD system. Primary outcome of the study is CAPD peritonitis rate and transfer set contamination rate between the two groups. The secondary outcomes are overall health conditions measured by two sets of standardized and reliable questionnaires: The short-form General Health Questionnaire (SF-36, Chinese version) and Depressive Anxiety Stress Scales (DASS-21, Chinese version).

[May refer to sessions of "Outcome measures" and "Eligibility" for details]

ELIGIBILITY:
Inclusion Criteria:

* Newly commenced CAPD patient in QEH
* Chose Ultrabag as PD system
* Planned to perform CAPD bag exchange by own
* Being assessed and categorized as "High to Moderate Readiness" to perform CAPD by Occupational Therapist
* Able to understand Cantonese, Putonghua or English

Exclusion Criteria:

* Severe cognitively impaired, aphasia, or suffer from psychiatric illness (e.g., unable to communicate effectively and understand the bag exchange procedure)
* old age home residents
* suffer from acute illness other than uremic syndromes requiring frequent hospital admission in the past 1 year (> 3 episodes with hospital stay over 1 week)
* adopt other assistive device in CAPD bag exchange procedure prescribed by Occupational Therapist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Peritonitis Rate | From the date of randomization until the end of the study (1 year post-training follow-up) or date of drop-out (e.g., peritonitis, death, refusal to participate in the study... etc) whichever came earlier, assessed up to 36 months.
  Peritonitis rate, in episodes per patient-year, as calculated by record of episodes of peritonitis and total number of patient months. Stratification of this outcome measure into intervention/ control arm for survival analysis could represent device safety.

SECONDARY OUTCOMES:
Health Scores | Through study completion, an average of 9 months at 4 timepoints: A0 (baseline), A1 (up to 1 month from recruitment to scheduled training session, and recorded at the end of the 1-week training), A2 (4-month post-training), A3 (8-month post-training).
  Health Scores as measured by short-form General Health Questionnaire (SF-36, Chinese version) which consisted of i) physical functioning, ii) role limitations due to physical health, iii) role limitations due to emotional problems, iv) energy/ fatigue, v) emotional well-being, vi) social functioning, vii) pain, and viii) general health with scores ranging from 0 (the worst) to 100 (the best).
Depressive Level | Through study completion, an average of 9 months at 4 timepoints: A0 (baseline), A1 (up to 1 month from recruitment to scheduled training session, and recorded at the end of the 1-week training), A2 (4-month post-training), A3 (8-month post-training).
  Depressive Level as assessed by the short-form Depressive Anxiety Stress Scales (DASS-21, Chinese version). Of 21 questions in DASS-21, 7 were extracted to calculate a sub-total score of the depression level, ranging from 0 to 21 (Normal = 0 - 4; Mild = 5 - 6; Moderate = 7 - 10; Severe = 11 - 13; Extremely Severe = 14 - 21).
Anxiety Level | Through study completion, an average of 9 months at 4 timepoints: A0 (baseline), A1 (up to 1 month from recruitment to scheduled training session, and recorded at the end of the 1-week training), A2 (4-month post-training), A3 (8-month post-training).
  Anxiety Level as assessed by the short-form Depressive Anxiety Stress Scales (DASS-21, Chinese version). Of 21 questions in DASS-21, 7 were extracted to calculate a sub-total score of the anxiety level, ranging from 0 to 21 (Normal = 0 - 3; Mild = 4 - 5; Moderate = 6 - 7; Severe = 8 - 9; Extremely Severe = 10 - 21).
Stress Level | Through study completion, an average of 9 months at 4 timepoints: A0 (baseline), A1 (up to 1 month from recruitment to scheduled training session, and recorded at the end of the 1-week training), A2 (4-month post-training), A3 (8-month post-training).
  Stress Level as assessed by the short-form Depressive Anxiety Stress Scales (DASS-21, Chinese version). Of 21 questions in DASS-21, 7 were extracted to calculate a sub-total score of the stress level, ranging from 0 to 21 (Normal = 0 - 7; Mild = 8 - 9; Moderate = 10 - 12; Severe = 13 - 16; Extremely Severe = 17 - 21).

OTHER OUTCOMES:
Basic Knowledge Acquisition | Through the timepoint of training completion, an average of 5 weeks at 1 timepoint: A1 (at the end of the 1-week training following recruitment and scheduling time up to 1 month).
  Basic knowledge acquisition level as assessed by Knowledge Evaluation Index (KEI), a verbal exam to evaluate the degree to which participants acquire renal disease related knowledge, CAPD complications and exit site care on cognitive domain. KEI scores ranged from 0 to 100% (full mark; pass at 50%).
CAPD Performance | Through the timepoint of training completion, an average of 5 weeks at 1 timepoint: A1 (at the end of the 1-week training following recruitment and scheduling time up to 1 month).
  CAPD-specific skills acquisition as assessed by a practical summative assessment which evaluates hands-on skill acquisition of participants at the end of the training. Either Pass (perform entire procedures in correct order by self) or Fail (unable to complete all steps in correct order) will be determined on assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Carina HO, APN(Renal), Principal Investigator — Renal Unit, Queen Elizabeth Hospital
Locations (1):
- Renal Unit, Department of Medicine, QEH, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hsieh YP, Wang SC, Chang CC, Wen YK, Chiu PF, Yang Y. The negative impact of early peritonitis on continuous ambulatory peritoneal dialysis patients. Perit Dial Int. 2014 Sep-Oct;34(6):627-35. doi: 10.3747/pdi.2013.00024. Epub 2014 Feb 4. PMID 24497590
- [Background] Lam, E T P, Lam, C L K, Lo, Lo, YC Yvonne, Gandek, B. (2008). Psychometrics and population norm of the Chinese (HK) SF-36 Health Survey_Version 2, HK Pract, 30, 189-197
- [Background] Lee, A., Koo, J., Wan, S.H., Hui, Y. H., Wong, S. H. & Chan, K. H. (2018). Application of 3D Printing Technology in Fabrication of Renal Device for Self-Continuous Ambulatory Peritoneal Dialysis-A Pilot Study. HA Convention 2018.
- [Background] Li PK, Szeto CC, Piraino B, de Arteaga J, Fan S, Figueiredo AE, Fish DN, Goffin E, Kim YL, Salzer W, Struijk DG, Teitelbaum I, Johnson DW. ISPD Peritonitis Recommendations: 2016 Update on Prevention and Treatment. Perit Dial Int. 2016 Sep 10;36(5):481-508. doi: 10.3747/pdi.2016.00078. Epub 2016 Jun 9. No abstract available. PMID 27282851
- [Background] Moussa, M.T., Lovibond, P.F. & Laube, R. (2001). Psychometric properties of a Chinese version of the short Depression Anxiety Stress Scales (DASS21). Report for New South Wales Transcultural Mental Health Centre, Cumberland Hospital, Sydney; Available at: http://www2.psy.unsw.edu.au/groups/dass/Chinese/tmhc.htm
- [Background] Szeto CC, Li PK. Peritoneal Dialysis-Associated Peritonitis. Clin J Am Soc Nephrol. 2019 Jul 5;14(7):1100-1105. doi: 10.2215/CJN.14631218. Epub 2019 May 8. PMID 31068338